CLINICAL TRIAL: NCT06987396
Title: Clinical Investigation to Assess the Effect of Betaglucan Administration in HPV Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitae Health Innovation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VITAE HEALTH INNOVATION S.L.
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: HPV
Keywords: HPV; Betaglucans; Immunity; RNA

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: RNA and DNA PCR tests were performed by a blinded external laboratory
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated group with 1000 mg oral Betaglucans (Immunovita) (Experimental)
  Interventions: Dietary Supplement: 1000 mg Betaglucans (daily)
- Control group without treatment (active surveillance) (No Intervention)

INTERVENTIONS:
Dietary Supplement: 1000 mg Betaglucans (daily) — Patients in the experimental group receive betaglucans supplement in capsule form, administered orally
  Arms: Treated group with 1000 mg oral Betaglucans (Immunovita)

SUMMARY:
Randomised, controlled clinical study to assess the efficacy and tolerability of an oral supplementation of 1000 mg daily of Betaglucans in the evolution of patients with Human Papilloma Virus (HPV). The improvement is measured by DNA PCR test, cytology and a specific RNA test.

ELIGIBILITY:
Inclusion Criteria:

* Women over 30 years old, whether or not they have been vaccinated against HPV
* Patients attending a visit with a routine cytological result of ASCUS or lSIL, or a normal result with a positive HPV test, no more than 3 months prior to be enrolled
* Patients who freely provide written informed consent
* Patients with a positive DNA PCR test

Exclusion Criteria:

* Patients who are participating in another clinical study about the same or different condition within the 30 days prior to inclusion.
* Any subject who, in the investigator's opinion, is unable to follow instructions or properly comply with the treatment.
* Subjects who do not provide written informed consent to participate in the study.
* Patients who are receiving any of the prohibited drugs or supplements, and for whom withdrawal of these medications/products is expected to pose a significant issue.
* Pregnant or breastfeeding women.
* Transplanted patients and/or patients taking immunosuppressive medication.
* Patients with autoimmune diseases.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 80 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
RNA PCR Test result | From enrollment to the end of treatment at 6 months

SECONDARY OUTCOMES:
DNA PCR Test result | From enrollment to the end of treatment at 6 months
Citology Test result | From enrollment to the end of treatment at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gynaecology Department, Medical Service Ishtar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No